CLINICAL TRIAL: NCT00355810
Title: Lactobacillus Plantarum MF 1298 vs Placebo for Irritable Bowel Syndrome.
Brief Title: Probiotics for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Food Research (Unknown); Gilde (Other); Norwegian Foundation for Health and Rehabilitation (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REK 4.2005.2284
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Functional Gastrointestinal Disorders; Irritable Bowel Syndrome
Keywords: Probiotics
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo followed by probiotic (Experimental): placebo, then washout period, then Lactobacillus plantarum MF1298
  Interventions: Dietary Supplement: placebo followed by Lactobacillus plantarum MF 1298
- probiotic followed by placebo (Experimental): Lactobacillus plantarum MF1298, then washout period, then placebo
  Interventions: Dietary Supplement: Lactobacillus plantarum MF1298 followed by placebo

INTERVENTIONS:
Dietary Supplement: placebo followed by Lactobacillus plantarum MF 1298 — placebo during 3 weeks, washout period 4 weeks, Lactobacillus plantarum MF1298 during 3 weeks
  Other Names: probiotic
  Arms: placebo followed by probiotic
Dietary Supplement: Lactobacillus plantarum MF1298 followed by placebo — Lactobacillus plantarum MF1298 during 3 weeks, washout period 4 weeks, placebo during 3 weeks
  Other Names: probiotic
  Arms: probiotic followed by placebo

SUMMARY:
This randomised, double blind, cross-over study compares the effect (symptoms, fecal bacterial growth, gas production) of three weeks' treatment with lactobacillus plantarum MF 1298 with placebo in patients with irritable bowel syndrome. The results are related to dietary habits, food intolerance and food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome according to the Rome II criteria
* regular symptoms

Exclusion Criteria:

* Use of probiotics last three weeks
* pregnancy
* lactation
* co-existing other gastrointestinal disorders
* use of laxatives and antibiotics within last 5 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-01; Primary Completion 2006-04 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Satisfactory relief of abdominal symptoms | 11 weeks
  relief of symptoms recorded on diary cards

SECONDARY OUTCOMES:
Graded measurement of abdominal symptoms | 11 weeks
  IBS sum score
Fecal bacterial count | 11 weeks
Abdominal gas | 11 weeks
Immunological parameters | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Per G Farup, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Innlandet Hospital HF, Gjøvik, Oppland, Norway

REFERENCES:
- [Result] Ligaarden SC, Axelsson L, Naterstad K, Lydersen S, Farup PG. A candidate probiotic with unfavourable effects in subjects with irritable bowel syndrome: a randomised controlled trial. BMC Gastroenterol. 2010 Feb 10;10:16. doi: 10.1186/1471-230X-10-16. PMID 20144246
- [Result] Farup PG, Jacobsen M, Ligaarden SC, Rudi K. Probiotics, symptoms, and gut microbiota: what are the relations? A randomized controlled trial in subjects with irritable bowel syndrome. Gastroenterol Res Pract. 2012;2012:214102. doi: 10.1155/2012/214102. Epub 2012 Jul 31. PMID 22899904